CLINICAL TRIAL: NCT06573671
Title: Histiocytosis in Injecting Drug Users
Status: Enrolling by invitation | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Oulu (Other); University of Turku (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Other Study IDs: R20105
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Histiocytosis
Keywords: intravenous; drug abuse; polyvinylpyrrolidone; PVP
MeSH Terms: conditions — Histiocytosis; Substance-Related Disorders | interventions — Microscopy, Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Biospecimen Retention: Samples With DNA — Blood samples for RNA analyses (transcriptomics) Coded patient tissue biopsies containing histiocytosis Healthy tissue and other histiocytosis tissues from biobank(s) serve as controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Injecting drug induced histiocytosis: No intervention
  Interventions: Diagnostic Test: Chitotriosidase; Diagnostic Test: Mass spectrometry; Diagnostic Test: scanning electron microscope with energy-dispersive X-ray spectroscopy; Diagnostic Test: Fluorescence microscopy; Diagnostic Test: Transcriptomics

INTERVENTIONS:
Diagnostic Test: Chitotriosidase — The amount of patients with increased chitotriosidase, and the extent of elevation of chitotriosidase
Diagnostic Test: Mass spectrometry — to show polyvinylpyrrolidone presence in histiocytes of injecting drug users compared to controls
Diagnostic Test: scanning electron microscope with energy-dispersive X-ray spectroscopy — to show polyvinylpyrrolidone presence in histiocytes of injecting drug users compared to controls
Diagnostic Test: Fluorescence microscopy — to show polyvinylpyrrolidone presence in histiocytes of injecting drug users compared to controls
Diagnostic Test: Transcriptomics — To describe pathologic signals of polyvinylpyrrolidone-exposed in vitro histiocytes of injecting drug users compared to control samples

SUMMARY:
The goal of this observational study is to describe a new disease condition of histiocytosis related to injecting drug use, its preconditions, symptoms, signs, findings, and prognosis in a detailed and systematic patient series in one referral center. The main question[s] it aims to answer are:

* to find specific histologic features in different tissues to help the differential diagnosis from other histiocytoses
* to describe the value of chitotriosidase activity to screen this condition
* to describe the value of various tissue biopsies in confirming the diagnosis
* to describe the nature of polyvinylpyrrolidone accumulation in tissue macrophages by novel special microscopic techniques
* to find new tandem mass spectrometry methodology to prove polyvinylpyrrolidone accumulation in macrophages
* to show that polyvinylpyrrolidone treatment activates macrophages to histiocytes and causes povidone accumulation within the cells in in vitro experiments
* to evaluate the pathology of macrophage activation to histiocytes by transcriptomics

The patient history will be collected from the data produced by follow-up of cases followed up in a single center. A subgroup of participants will be given an opportunity to sign informed consent to give access to/donate blood and tissue samples to search for techniques to prove polyvinylpyrrolidone storage within histiocytes, and to search for transcriptomics signal(s) in histiocytes.

Researchers will compare blood and tissue samples from the biobank as controls.

DETAILED DESCRIPTION:
Comprehensive patient data (disease history, findings, complications, laboratory findings, histopathology, and imaging) will be obtained from patient records of a single university hospital. Coded histiocytosis-positive tissue samples will be compared to biobank samples from corresponding tissues from healthy and other histiocytosis tissue samples to show polyvinylpyrrolidone storage with novel methodologies.

In addition, if a study participant who is followed up clinically, signs informed consent, monocytes are separated from a blood sample, differentiated to macrophages, and exposed to polyvinylpyrrolidone. Various novel methods will be utilized to explore polyvinylpyrrolidone within histiocytes.

ELIGIBILITY:
Inclusion Criteria:

* All identified adult patients in our records with a history of injecting drug use by dissolving tablets containing polyvinylpyrrolidone and (suspected) PVP-histiocytosis

Exclusion Criteria:

* Other histiocytosis diagnosed by tissue samples and clinical information

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitting to intravenous use of dissolved tablets (indicated for oral use) containing polyvinylpyrrolidone (PVP30) and positive tissue sample in any tissue biopsy compatible with features of histiocytosis caused by PVP30
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of disease manifestations | 10 years
  To describe phenotype

SECONDARY OUTCOMES:
Frequency of elevated chitotriosidase activity | 10 years
  Is chitotriosidase activity associated with polyvinylpyrrolidone histiocytosis
Mortality | 10 years
  Mortality
Microscopic fluorescence positive tissue | 10 years
  Search for specific polyvinylpyrrolidone fluorescence signal
Scanning electron microscope with energy-dispersive X-ray spectroscopy | 10 years
  search for specific polyvinylpyrrolidone signal within cells
Pyrolysis mass spectrometry | 10 years
  search for specific polyvinylpyrrolidone signal within cells
Transcriptomics analysis | 10 years
  Search for immunologic pathway-specific abnormalities to guide treatment in cases compared with controls

CONTACTS AND LOCATIONS:
Overall Officials: Pasi I Nevalainen, MD, PhD, Principal Investigator — Senior consultant
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
Study data can only be acquired by proper inquiry to the national authority Findata by law